CLINICAL TRIAL: NCT00630435
Title: An Open-Label, Single-Dose, Randomized, 4-Period, Crossover, Bioequivalence Study of 3 New Formulations of Premarin® /MPA 0.625 mg/2.5 mg Compared With Reference Formulation of Premarin®/MPA in Healthy Postmenopausal Women
Brief Title: Study Comparing 3 New Formulations of Premarin® 0.625 mg/MPA 2.5 mg With a Reference Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 0713E1-1137
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Menopause
Keywords: Premarin®

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Premarin®/MPA formulation A
- 2 (Experimental)
  Interventions: Drug: Premarin®/MPA formulation B
- 3 (Experimental)
  Interventions: Drug: Premarin®/MPA formulation C
- 4 (Active Comparator)
  Interventions: Drug: Premarin®/MPA currently marketed product

INTERVENTIONS:
Drug: Premarin®/MPA formulation A
  Arms: 1
Drug: Premarin®/MPA formulation B
  Arms: 2
Drug: Premarin®/MPA formulation C
  Arms: 3
Drug: Premarin®/MPA currently marketed product
  Arms: 4

SUMMARY:
The purpose of this trial is to determine the equivalence of 3 new formulations of a Premarin®/medroxyprogesterone acetate (MPA) combination tablet to the currently marketed dosage form (Prempro® [TM]). This study will be performed in healthy postmenopausal women. Each subject will participate in the study for approximately 14 weeks, including a screening evaluation within 3 weeks before the study, and four, 6-day, 5-night inpatient periods with at least a 21-day washout interval between each dose administration.

ELIGIBILITY:
Inclusion

1. Healthy postmenopausal women aged 35 to 70.
2. Body mass index of 18 to 35 kg/m2, weight must be at least 50 kg.
3. Nonsmoker or smoker of fewer than 10 cigarettes/day.

Exclusion

1. History or presence of hypertension (>139 mm Hg systolic or >89 mm Hg diastolic). Can take up to 2 antihypertensive medications to keep blood pressure under control.
2. History within 1 year of study day 1 of alcohol or drug abuse.
3. Use of any investigational drug within 30 days before study day 1.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of Premarin® and medroxyprogesterone acetate between test and currently marketed formulations | 14 weeks

SECONDARY OUTCOMES:
No secondary outcome | No time frame

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer